CLINICAL TRIAL: NCT01985789
Title: The Effect of Antihistamines on Methacholine Challenge Testing in Asthma Patients
Brief Title: Anti-histamines and Methacholine Challenges.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Don Cockcroft (Other)
Responsible Party: Sponsor-Investigator, Don Cockcroft, Professor, University of Saskatchewan
Organization: University of Saskatchewan (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Diagnostic
Other Study IDs: PHPY2013/14
Record Dates: First submitted 2013-10-31; First posted 2013-11-15 (Estimated); Last update posted 2015-04-08 (Estimated); Status verified 2015-04

CONDITIONS: Asthma
Keywords: airway hyperresponsiveness
MeSH Terms: conditions — Asthma; Respiratory Hypersensitivity | interventions — Diphenhydramine; Cetirizine; desloratadine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- diphenhydramine (Active Comparator): 50mg dose given as two 25mg capsules
  Interventions: Drug: Diphenhydramine
- cetirizine (Active Comparator): 10mg dose given as 1 10mg capsule and 1 placebo capsule
  Interventions: Drug: cetirizine
- desloratadine (Active Comparator): 5mg dose given as 1 5mg capsule and 1 placebo capsule
  Interventions: Drug: desloratadine
- placebo (Placebo Comparator): given as 2 placebo capsules
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Diphenhydramine
  Arms: diphenhydramine
Drug: cetirizine
  Arms: cetirizine
Drug: desloratadine
  Arms: desloratadine
Drug: placebo
  Arms: placebo

SUMMARY:
The asthmatic airway is identified and studied using inhaled agents such as histamine and methacholine. The use of antihistamines prior to the test will inhibit the test result if histamine is used to cause airway constriction. If using methacholine, this may also be true depending on whether old (e.g. benadryl) or new (e.g. desloratadine) antihistamines are used. This study will look at the effect of old and new antihistamines on inhaled methacholine challenge response in individuals with mild asthma.

ELIGIBILITY:
Inclusion Criteria:

* Baseline forced expiratory volume in 1s (FEV1) of 70% or more of predicted
* Methacholine provocative concentration causing a 20% fall in FEV1 16mg/ml or less
* No respiratory infection or change in allergen exposure for 4 weeks prior to screening and throughout the study
* No significant medical co-morbidities
* allergy

Exclusion Criteria:

* pregnant or breastfeeding females
* unable to withhold antihistamines, anticholinergics, long acting bronchodilators and combination therapies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-11; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
change in methacholine pc20 | change from baseline (pre dose) at 2 hours (post dose)

CONTACTS AND LOCATIONS:
Overall Officials: Donald W Cockcroft, MD, Principal Investigator — University of Saskatchewan, Department of Medicine, Division of Respirology, Critical Care and Sleep Medicine
Locations (1):
- University of Saskatchewan, Saskatoon, Saskatchewan, Canada